CLINICAL TRIAL: NCT06049095
Title: A Sequential, Randomized, Double-Blind, Placebo-Controlled, Phase 1 Single and Multiple Ascending Dose Study of LTG-001 Administered Orally of Intravenously to Evaluate the Safety, Tolerability, and Pharmacokinetics in Healthy Male and Female Participants 18 to 55 Years of Age
Brief Title: A Phase 1 Single and Multiple Ascending Dose Study of LTG-001 Administered Orally in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Latigo Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LTG-001-001
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LTG-001 (Experimental): Part A: Single-Ascending dose cohorts; relative bioavailability; food effect; Part B: Multiple-ascending dose cohorts
  Interventions: Drug: LTG-001
- Placebo (Placebo Comparator): Part A: Single-Ascending dose cohorts; Part B: Multiple-ascending dose cohorts
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LTG-001 — Oral doses
  Arms: LTG-001
Drug: Placebo — Oral doses
  Arms: Placebo

SUMMARY:
This is a sequential, randomized, double-blind, placebo-controlled Phase 1 single (SAD) and multiple (MAD) ascending dose study to evaluate the safety, tolerability, and pharmacokinetics (PK) of orally or intravenously administered LTG-001 in healthy male and female participants

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 18 to 55 years, inclusive, at the time of signing the informed consent.
* Overtly healthy with no clinically relevant abnormalities based on the medical history, physical examinations, clinical laboratory evaluations, and 12-lead ECG that, in the opinion of the investigator, would affect participant safety.
* Body mass index (BMI) within the range of 18-32 kg/m2 (inclusive).

Exclusion Criteria:

* Inability to take oral medications or gastrointestinal abnormalities potentially impacting absorption
* Clinically significant cardiovascular, hematological, renal, hepatic, pulmonary, endocrine, gastrointestinal, immunological, dermatological, neurological, or psychiatric disease which could interfere with, or the treatment for which might interfere with, the conduct of the study or which would, in the opinion of the investigator, unacceptably increase the participant's risk by participating in the study
* Past or current history or evidence of alcohol abuse and/or dependence on recreational drug use
* Donation of over 500 mL blood ≤ 3 months prior to start of participation
* Has known psychiatric disorders that would interfere with the cooperation with the requirements of the study
* Participant is under legal custodianship.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 204 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2026-04-28 (Estimated); Study Completion 2026-04-28 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of single and multiple ascending oral doses, relative bioavailability and food effect of LTG-001 in healthy subjects | Up to 10 days of dosing
  Incidence, severity, seriousness, and causality of treatment-emergent adverse events (TEAEs)
Absolute Bioavailability of LTG-001 Following Oral and Intravenous Administration | from admission to completion in the study (35 days)
  Absolute bioavailability of LTG-001 will be assessed by comparing systemic exposure following a single oral tablet dose and a single intravenous dose.
Safety and Tolerability of Intravenous LTG-001 | From first intravenous dose through end of study (up to 14 days following intravenous dosing)
  Safety and tolerability of intravenous LTG-001 will be assessed by the number of participants with treatment-emergent adverse events (TEAEs), changes in clinical laboratory parameters, vital signs, electrocardiograms (ECGs), physical examination findings, and infusion site reactions following intravenous administration.

SECONDARY OUTCOMES:
To further characterize the PK of LTG-001 in healthy participants | Up to 10 days of dosing
  Cmax
To further characterize the PK of LTG-001 in healthy participants | Up to 10 days of dosing
  Area under the concentration curve from 0 to last (AUC0-last)
To further characterize the PK of LTG-001 in healthy participants | Up to 10 days of dosing
  Area under the concentration curve from 0 to infinity (AUC0-inf)
To further characterize the PK of LTG-001 in healthy participants | Up to 10 days of dosing
  Time of the maximum observed plasma concentration (tmax)
To further characterize the PK of LTG-001 in healthy participants | Up to 10 days of dosing
  Elimination rate constant (λz)
To further characterize the PK of LTG-001 in healthy participants | Up to 10 days of dosing
  Terminal elimination half-life (t1⁄2)
To further characterize the PK of LTG-001 in healthy participants | Up to 10 days of dosing
  Concentration at 12 hours (C12)
To further characterize the PK of LTG-001 in healthy participants | Up to 10 days of dosing
  Oral clearance (CL/F)
To further characterize the PK of LTG-001 in healthy participants | Up to 10 days of dosing
  Oral apparent volume of distribution (Vz/F)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Unit, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No